CLINICAL TRIAL: NCT04617912
Title: Evaluation of Long-Axial Field-of-View Positron Emission Tomography (PET) Scanner
Brief Title: PennPET Explorer Scanner Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 843546
Record Dates: First submitted 2020-09-14; First posted 2020-11-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PennPET Explorer (Experimental): All subjects will be scanned in the CT scanner and then the scanner bed will be moved into position in the PennPET Explorer for initiation of the PET scan. For all PET scans a radioactive imaging drug is used.
  The radiotracer injection may be performed according to one of the following scenarios:
  1. As part of a clinical standard-of-care (SOC) PET/CT or PET/MRI scan (using an FDA-approved radiotracer; the PennPET Explorer cannot yet accommodate a study that requires a commercially available 510(k)-approved instrument for clinical results, subjects in this group will be scanned on both a commercial instrument (PET/CT or PET.MRI) and the PennPET Explorer),
  2. As part of another research study (using either an FDA-approved radiotracer or an investigational radiotracer),
  3. As a research injection designed specifically to utilize the PennPET Explorer (using an FDA-approved radiotracer).
  Interventions: Device: Long AFOV PennPET Explorer

INTERVENTIONS:
Device: Long AFOV PennPET Explorer — A long-axial field-of-view (LAFOV) time-of-flight PET scanner, developed at the University of Pennsylvania, being tested for real-world applications.

SUMMARY:
Positron Emission Tomography (PET) is a procedure that uses a special type of machine to take pictures of the inside of the body after a radioactive drug is administered. The radioactive drug that is used for this study may be an FDA approved imaging drug or may be used as an investigational imaging drug as part of another study for which participants are taking part. PET using various radiotracers is useful for the diagnosis of various diseases, including cancer, brain diseases, infection, and heart or lung disease.

The purpose of this study is to test a research PET machine called the PennPET Explorer long-axial field-of-view scanner. This research PET machine can image a larger section of the body than the current clinical PET scanners, allowing most of the body to be imaged at one time. This scanner is still an investigational device and is being tested in this study to collect more information about how best to use this type of whole body scanner.

DETAILED DESCRIPTION:
The PennPET Explorer is a multiring system with a long AFOV that is scalable and comprised of multiple 22.9 cm long ring segments, each with 18 detector modules based on a commercial digital silicon photomultiplier. Initial testing data on a prototype 3-ring-segment instrument with an active 64-cm AFOV has been collected and published by Karp et al., and Pantel et al., [Karp 2020, Pantel 2020], validating the system design and demonstrating its initial performance.

In the last two decades, commercial PET scanner performance has improved dramatically with CT-based attenuation correction 1, the use of lutetium oxyorthosilicate or lutetium-yttrium oxyorthosilicate scintillators, time-of-flight reconstruction 2-5, and, most recently, silicon photomultiplier (SiPM)-based time-of-flight detectors 2,6. However, the AFOV has not grown; it remains 16-26 cm for the newest commercial SiPM-based scanners 7,8. This choice is due mainly to scintillator and SiPM photosensor costs and the prevalence of clinical 18F-FDG scanning focused on measuring lesion SUV when the uptake is assumed to be at steady state, typically at 60 min after injection. The newest commercial instruments perform an 18F-FDG whole-body survey (skull-base to mid-thigh) with excellent diagnostic quality in 10-20 min using bed translation.

The motivation for a LAFOV PET system is to use its high sensitivity to enhance clinical performance and to enable research applications. Clinically, a LAFOV system could enable faster imaging, imaging with lower injected activities, or a combination of the two. Research applications include delayed imaging, improving quantification for kinetic modeling, and applications requiring simultaneous measurement of multiple organ systems 9,10. It is unknown whether such a system would primarily be used for clinical or research applications. The investigators developed the PennPET Explorer whole-body imager to support both applications. Performance measurements were taken on the prototype 3-ring-segment system to optimize the hardware and software acquisition and reconstruction, as well as to demonstrate the capabilities of the PennPET Explorer. The investigators are operating with a total of 6 ring-segments which will give an active 140 cm AFOV. This will allow whole-body imaging in one bed position for most adults.

In the evaluation of a new instrument, human studies are essential to establish the real-world performance beyond phantom studies, as well as to test and optimize data acquisition and reconstruction. To date 11 human studies have been imaged on the prototype scanner under IRB 809476. This instrument was determined by the FDA to meet the definition of a nonsignificant risk (NSR) device and is therefore subject only to abbreviated IDE requirements. Once the additional ring-segments have been added to the instrument, the investigators plan to continue testing this scanner in human subjects under this ongoing open-ended protocol. The investigators will continue to work towards optimizing performance and data acquisition until such time as this device receives full FDA 510(k) approval.

This protocol is designed to test the PennPET Explorer instrument with its final AFOV of 140 cm. PET imaging involves the administration of a radioactive imaging drug that emits positrons which are detected by the scanner and used to form the images. For the purposes of this protocol, the administered radioactive imaging drug (tracer) will vary; it may be an FDA-approved radiotracer or an experimental radiotracer that is used under an IND. If the radiotracer used is under an IND, then the administration of the radiotracer will be done under the purview of a separate protocol for which the subject has been separately consented. This protocol and the corresponding ICF involves consent only for being scanned on the investigational scanner and does not pertain to the administration of an investigational radiopharmaceutical.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, at least 18 years of age
* Participants or study partner must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures. Subjects who are unable to provide consent must have a legally authorized representative or designated "study partner" who can provide consent on their behalf.

Exclusion Criteria:

* Inability to tolerate imaging procedure in the opinion of an investigator.
* Serious or unstable medical or psychological conditions or lack of mobility that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Image Performance of the LAFOV PennPET Explorer | Through study completion, an average of 1 year.
  Noise behavior, structural detail and local contrast will be combined to report overall image quality using a numerical scale (1 = poor image quality, 5 = superior image quality).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No